CLINICAL TRIAL: NCT06736990
Title: A Randomized Double-Blind Trial to Evaluate the Efficacy and Safety of CAL101 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Phase 2 Study of CAL101 in Patients With Idiopathic Pulmonary Fibrosis
Acronym: AURORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Calluna Pharma AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAL101-201; 2024-518339-12-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-16; First posted 2024-12-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — idelalisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAL101 (Experimental)
  Interventions: Drug: CAL101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAL101 — Intravenous infusions of CAL101 every 4 weeks over 24 weeks
  Arms: CAL101
Drug: Placebo — Intravenous infusions of placebo every 4 weeks over 24 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the investigational drug CAL101 can help prevent further decline in lung function in adults with Idiopathic Pulmonary Fibrosis.

Researchers will compare CAL101 with placebo to compare change from baseline in forced vital capacity (FVC).

Participants will be randomly assigned to a study group that will receive an IV infusion of either the study medication or placebo about once a month for 6 months.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of CAL101 in participants with IPF, either as standalone treatment or in addition to currently approved antifibrotic treatments..

The study will consist of a 28-days Screening Period, intravenous (IV) infusions of CAL101 or placebo once every 4 weeks over 24 weeks, and a 16 week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 years of age
* Diagnosis of IPF supported by centrally read chest high-resolution computed tomography
* Definite or probable usual interstitial pneumonia (UIP) pattern on chest high-resolution computed tomography (HRCT) performed within 12 months of screening, confirmed by central review (if an evaluable HRCT < 12 months is not available, the baseline HRCT will be used to determine eligibility).
* FVC ≥ 45% of predicted (at Screening).
* Diffusing capacity of the lung for carbon monoxide (DLCO) ≥ 25% predicted.
* Forced expiratory volume in 1 second (FEV1)/FVC ≥ 0.70 at Screening or FEV1/FVC ≥ predicted value minus 0.10 (if predicted value according to the spirometry report at Screening is <0.80).
* Either stable dose with an approved antifibrotic for at least 8 weeks prior to screening or not treated with antifibrotics for at least 8 weeks prior to screening.

Exclusion Criteria:

* In the opinion of the Investigator, other clinically significant lung disease (e.g. asthma, emphysema, chronic obstructive pulmonary disease, cavitary or pleural diseases, clinically significant or treatment-requiring pulmonary hypertension) at screening.
* Interstitial lung disease (ILD) other than IPF (including, but not limited to, connective tissue diseases, vasculitis).
* Acute IPF exacerbation within 16 weeks prior to screening and/or during the screening period (investigator-determined).
* Lower respiratory tract infection requiring antibiotics within 4 weeks prior to screening and/or during the screening period.
* Evidence of impaired kidney function, unstable cardiovascular disease, moderate or severe hepatic impairment or any significant disease or condition other than IPF which may interfere with trial procedures or interpretation of trial results, or cause concern regarding the patient's ability to participate in the trial or any medical condition which could lead to a life expectancy < 12months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in forced vital capacity (FVC) compared to placebo | 28 weeks

CONTACTS AND LOCATIONS:
Locations (54):
- United States (9):
  - Keck School of Medicine at USC, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Y & L Advance Health Care, Inc. d/b/a Elite Clinical Research, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Pulmonix, LLC, Greensboro, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Utah Health, Salt Lake City, Utah
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (5):
  - AP-HP Hopital Avicenne, Bobigny
  - AP-HP Hopital Europeen Georges Pompidou, Paris
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - CHU de Toulouse - Hopital Larrey, Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours
- Italy (7):
  - Azienda Ospedale - Università Padova, Padua, PD
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma, RM
  - Azienda Ospedaliero Universitaria Senese, Siena, SI
  - Azienda sanitaria universitaria Giuliano Isontina (ASU GI) - Ospedale di Cattinara, Trieste, TS
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - AORN - Ospedali dei Colli - Ospedale V. Monaldi, Napoli
  - Istituto Clinico Humanitas - Pneumologia 1, Rozzano
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - St. Antonius Ziekenhuis - Locatie Nieuwegein, Nieuwegein, Utrecht
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Rikshospitalet, Oslo
- Romania (4):
  - Spitalul Clinic de Pneumoftiziologie ''Leon Daniello'', Cluj-Napoca, Cluj
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie ''Victor Babes'' Craiova, Craiova, Dolj
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie dr. Victor Babes Timisoara, Timișoara, Timiș County
  - Institutul de Pneumoftiziologie Marius Nasta, Bucharest
- South Korea (5):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- Turkey (Türkiye) (3):
  - University of Health Sciences Gulhane Faculty of Medicine, Ankara
  - Uludag University Medical Faculty, Bursa
  - Ege University Medical Faculty Hospital, Izmir
- United Kingdom (9):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - NHS Lothian, Edinburgh Royal Infirmary, Edinburgh
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Brompton Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borchert SV, Hallen J, Hussain RI, Holyer I, Troelsen JT, Klingelhofer J. Development of CAL101-a humanized monoclonal antibody targeting S100A4 to inhibit proinflammatory and profibrotic signaling. J Pharmacol Exp Ther. 2025 Nov;392(11):103722. doi: 10.1016/j.jpet.2025.103722. Epub 2025 Sep 24. PMID 41124966